CLINICAL TRIAL: NCT00291980
Title: A Phase III, Multicentric, Multinational, Controlled, Randomised, Open Study Comparing the Immunogenicity, Reactogenicity and Safety of Henogen's New Adjuvanted Hepatitis B Vaccine, HB-AS02V, to That of Aventis Pasteur MSD's Hepatitis B Vaccine, HBVAXPRO® , Administered as a Booster Dose in Pre-Dialysis, Peritoneal Dialysis and Haemodialysis Subjects (³ 15 Years of Age) Who Previously Responded to Hepatitis B Primary Vaccination But Have Lost Antibody.
Brief Title: A Study to Compare the Immune Response and Safety Elicited by Henogen's Adjuvanted Hepatitis B Vaccine Compared to Aventis Pasteur MSD's Hepatitis B Vaccine in Pre-Dialysis and Dialysis Patients Who Responded to Previous Hepatitis B Vaccination But Lost Antibody.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Henogen (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sophie Houard CSO, Henogen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HN018/HBV-004 (105754); NCT00739804 (obsolete NCT alias)
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2008-08-28 (Estimated); Status verified 2008-08

CONDITIONS: Hepatitis B
Keywords: Dialysis; Pre-dialysis; Hepatitis B vaccine; Prophylaxis hepatitis B infection
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): HB-AS02V vaccine
  Interventions: Biological: HB-AS02V vaccine
- 2 (Active Comparator): HBVAXPRO vaccine
  Interventions: Biological: HBVAXPRO vaccine

INTERVENTIONS:
Biological: HB-AS02V vaccine — HB-AS02V (20µg HBsAg) will be administered at Month 0
  Arms: 1
Biological: HBVAXPRO vaccine — HBVAXPRO vaccine (40µg HBsAg) will be administered at Month 0
  Arms: 2

SUMMARY:
The immune response of uraemic patients to hepatitis B vaccination is impaired compared to healthy subjects. After vaccination, anti-HBs peak antibody concentrations are reduced. As the persistence of anti-HBs is closely related to the initial anti-HBs peak, a more immunogenic vaccine, allowing higher antibody concentrations, would be a benefit for this population.

DETAILED DESCRIPTION:
Study participants will receive either Henogen's adjuvanted hepatitis B vaccine or Aventis Pasteur's hepatitis B vaccine. The study involves a total of 3 visits and blood samples will taken at each of these visits.

ELIGIBILITY:
Inclusion Criteria:

* Subjects whom the investigator believes that they can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits) should be enrolled in the study.
* A male or female subject 15 years of age or older at the time of the study entry.
* Written informed consent obtained from the subject/ subject's parents or guardians.
* Pre-dialysis patients, peritoneal dialysis patients and patients on haemodialysis. Pre-dialysis patients is defined as a subject with a documented creatinine clearance of les or equal to 30 ml/min.
* Seronegative for anti-HBc antibodies and for HBsAg at screening.
* Documented previous hepatitis B vaccination with one full primary course of licensed vaccine (the cumulative dose for primary vaccination is at least 160 mg of hepatitis B vaccine) with or without subsequent boosters. The last dose should have been administered at least three months before the planned dose of study vaccine in this study.
* Documented response to previous hepatitis B vaccination (i.e. anti-HBs antibody concentrations ³ 10 mIU/ml after primary vaccination or after booster/s with licensed vaccine), but for whom there is a loss of anti-HBs antibody concentrations below 10 mIU/ml at the time of inclusion into the study. Patients who have antibody concentrations below 50 mIU/ml at the time of inclusion will also be recruited provided that this antibody concentration is less than half of the highest documented antibody response achieved after primary vaccination or booster/s. The interval between the blood sample corresponding to the documented response and the hepatitis B vaccine dose received prior to this blood sample should be at least 25 days
* If the subject is female, she must be of non-childbearing potential, i.e., either surgically sterilized or one year post-menopausal; or, if of childbearing potential, she must be abstinent or have used medically-approved contraceptive precautions for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series.

Exclusion Criteria:

* Subjects who have participated in the HN014/HBV-001 or HN017/HBV-003 study
* Use of any investigational or non-registered drug or vaccine within 30 days preceding the study vaccine administration, or planned use during the study period.
* Use of any registered vaccine within 7 days preceding the study vaccine administration.
* History of hepatitis B infection.
* Known exposure to hepatitis B virus within six months.
* Use of immunoglobulins within six months preceding the first study vaccination.
* Immunosuppression caused by the administration of parenteral steroids or chemotherapy (oral steroids are allowed).
* Any confirmed or suspected human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* Acute disease at the time of enrolment. (Acute disease is defined as the presence of a moderate or severe illness with or without fever. All vaccines can be administered to persons with a minor illness such as diarrhoea, mild upper respiratory infection with or without low-grade febrile illness, i.e., oral/ axillary temperature < 37.5°C (or 37 °C in Czech Republic).
* Oral/axillary temperature equal or superior to 37.5 °C (or 37 °C in Czech Republic).
* Pregnant or lactating female

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2006-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Anti-HBs antibody geometric mean concentrations. | Month 0 and Month 1

SECONDARY OUTCOMES:
Seroprotection rates for all subjects | Months 0, 1
Seropositivity rates for all subjects | Month 0 and at Month 1
Percentage of subjects with anti-HBs antibody concentrations superior or equal to 100 mIU/ml for all subjects | Month 0 and at Month 1
Geometric Mean Concentration of anti-HBs antibodies for all subjects and for seropositive subjects | Month 0 and Month 1
Occurrence and intensity of solicited local signs and symptoms, relationship to vaccination of solicited general signs and symptoms during the 4-day follow-up after vaccination | Month 0
Occurrence, intensity and relationship to vaccination of unsolicited local and general signs and symptoms during the 31-day (Day 0 to Day 30) follow-up period after vaccination | Month 0
Occurrence, intensity and relationship to vaccination of all serious adverse events up to Month 1 | Month 0 to 1

CONTACTS AND LOCATIONS:
Overall Officials: Christian Tielemans, MD, PhD, Principal Investigator — ULB Hôpital Erasme Département de Néphrologie
Locations (28):
- Belgium (13):
  - O.L.Vrouwziekenhuis Aalst, Aalst
  - RHMS La Madeleine ATH, Ath
  - RHMS Clinique Louis Caty Baudour, Baudour
  - Cliniques universitaires Saint Luc, Brussels
  - CHU Brugmann (site V Horta) Service de néphrologie, Brussels
  - ULB Hôpital Erasme Département de Néphrologie, Brussels
  - CHU Hôpital civil de, Charleroi
  - UZ AntwerpenDienst nefrologie, Edegem
  - UZ Gent, Ghent
  - CHU Tivoli, La Louvière
  - UZ Gasthuisberg Leuven Nierziekten, Leuven
  - CHU Andre VESALE, Montigny-le-Tilleul
  - RHMS TournayService de néphrologie, Tournai
- Czechia (9):
  - Clinic of Gerontology and MetabolismDepartment of NephrologyUniversity HospitalSokolska, Hradec Králové
  - Hospital JihlavaVrchlického, Jihlava
  - Regional Hospital Liberec, Liberec
  - Dept. of NephrologyIII. Clinic of Internal DiseasesUniversity Hospital I.P.Pavlova, Olomouc
  - Infection Diseases and AIDS Treatment ClinicUniversity Hospital with Outpatient Clinic, Ostrava - Poruba
  - Fresenius Medical Care - DS, s.r.o.: PardubiceDialysis Unit Kyjevska, Pardubice
  - Fresenius Medical Care - DS Prague 4, Prague
  - Dept. of Internal Medicine StrahovSermirska 5, Prague
  - Fresenius Medical Care - DS, s.r.o.: SokolovDialysis Unit Slovenska, Sokolov
- Hungary (6):
  - University of Debrecen Medical and Science CenterI. Medical Clinic for Internal Diseases Nephrology Department, Debrecen
  - Markhot Ferenc County HospitalFresenius Dialysis Center Baktai, Eger
  - Vaszary Kolos HospitalFresenius Dialysis Center, Esztergom
  - Petz Aladár Teaching Hospital Vasvári, Győr
  - Hatvan Hospital Health Care ProviderFresenius Dialysis Center Hatvan ., Hatvan
  - Vas and Szombathely County Markusovszky Hospital, Szombathely